CLINICAL TRIAL: NCT05915611
Title: Evaluating the Effectiveness of a Combined Physical and Psychological Intervention in Carpal Tunnel Syndrome Patients With Nociplastic Pain: A Randomized Controlled Trial
Brief Title: Combined Physical and Psychological Intervention in Carpal Tunnel Syndrome Patients With Nociplastic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/CTS/120002023
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Carpal Tunnel Syndrome; Pain, Chronic
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain | interventions — Psychosocial Intervention; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive a twelve-week combined physical and psychological intervention.
  Interventions: Other: Combined physical and psychological intervention
- Control group (Active Comparator): Participants will receive a twelve-week of standard care of splinting, tendon and nerve gliding exercises.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Combined physical and psychological intervention — Physical therapy components will include splinting, tendon and nerve gliding exercises.
  Psychological components will include cognitive-behavioral therapy (CBT), delivered in individual sessions, targeting pain catastrophizing and fear of movement.
  Participants will attend 2 physical therapy sessions and one CBT session per week. for a period of 12 weeks
  Arms: Intervention group
Other: Standard care — Participants will be asked to wear a prefabricated wrist splint during the night and during strenuous activity. Also, they will receive tendon and nerve gliding exercises
  Arms: Control group

SUMMARY:
To assess the effectiveness of a combined physical and psychological intervention in reducing pain and improving function in carpal tunnel syndrome patients with nociplastic pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25-65 years
* Both sexes
* Diagnosis of carpal tunnel syndrome based on clinical examination and nerve conduction studies
* Presence of nociplastic pain as determined by the Central Sensitization Inventory (CSI) with a score ≥40
* Positive tinel and phalen sign.

Exclusion Criteria:

* Previous carpal tunnel release surgery
* Other musculoskeletal or neurological disorders affecting the upper extremity

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-27 (Estimated); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Pain intensity using the Numeric Pain Rating Scale (NPRS) | Changes in pain intensity at baseline, 6 weeks, 12 weeks.
Functional ability using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Changes in Functional ability at baseline, 6 weeks, 12 weeks.
Median nerve motor distal latency | Changes in Median nerve motor distal latency at baseline, 6 weeks, 12 weeks.
Median nerve sensory distal latency | Changes in Median nerve sensory distal latency at baseline, 6 weeks, 12 weeks.

SECONDARY OUTCOMES:
Pain catastrophizing using the Pain Catastrophizing Scale (PCS) | Changes in Pain Catastrophizing Scale (PCS) at baseline, 6 weeks, 12 weeks.
Fear of movement using the Tampa Scale for Kinesiophobia (TSK) | Changes in Tampa Scale for Kinesiophobia (TSK) at baseline, 6 weeks, 12 weeks.
Grip strength measured using a hand dynamometer | Changes in Grip strength at baseline, 6 weeks, 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No